CLINICAL TRIAL: NCT06480045
Title: Usage Of Artificial Intelligence-Integrated Usg In Application of Pectoral Block In Mastectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Çağla Yazar, MD, Principal investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA21/353
Record Dates: First submitted 2023-12-07; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasms
Keywords: mastectomy; pectoral nerve block; USG; artificial intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 70 patients with ASA I-II, between the ages of 18-75, who were scheduled for mastectomy surgery were included in the study. An anesthesiology resident under the supervision of senior anesthesiologist, performed a PECS II block with AI-integrated USG or conventional USG (Group AI-USG and Group USG) after randomization. Block was performed after induction of general anesthesia. Patient data in terms of hemodynamic changes in the intraoperative period, opioid consumption, and postoperatively hemodynamics, pain scores (VAS), postoperative opioid (tramadol administered with a patient-controlled analgesia pump) and, if necessary, rescue analgesic agent (non-steroidal antiinflammatory agent) consumption were monitored in the post-anesthesia care unit, and at postoperative 6., 12. and 24.hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group AI-USG (Active Comparator): performed a PECS II block with AI-integrated USG
  Interventions: Procedure: Performed PECS II block with AI integrated USG
- Group USG (Active Comparator): performed a PECS II block with conventional USG
  Interventions: Procedure: Performed PECS II block with conventional USG

INTERVENTIONS:
Procedure: Performed PECS II block with AI integrated USG — A 4-year anesthesiology resident, under the supervision of two senior anesthesiologists, performed a PECS II block with AI-integrated USG.
  Arms: Group AI-USG
Procedure: Performed PECS II block with conventional USG — A 4-year anesthesiology resident, under the supervision of two senior anesthesiologists, performed a PECS II block with conventional USG.
  Arms: Group USG

SUMMARY:
The investigator's goal in this study is to apply PECS II block, before starting surgery, by either conventional USG or artificial intelligence integrated USG to patients who will undergo mastectomy under general anesthesia to determine the effect of the block on hemodynamics and opioid consumption in the intraoperative period. Besides, the investigatorwanted to investigate the contribution of artificial intelligence integrated USG use in the success of a 4-year anesthesiology resident for imaging the injection site.

DETAILED DESCRIPTION:
After receiving the approval of the Clinical Research Ethics Committee of Başkent University (KA21/353), 70 patients with ASA I-II, between the ages of 18-75, who were scheduled for mastectomy surgery were included in the study. A 4. year anesthesiology resident under the supervision of two senior anesthesiologists, performed a PECS II block with AI-integrated USG or conventional USG (Group AI-USG and Group USG) after randomization. Although the resident had no experience with pectoral blocks, she had experience with the use of USG and regional anesthesia related to other trunk-area and peripheral blocks. The block was performed after induction of general anesthesia. Patient data in terms of hemodynamic changes in the intraoperative period, opioid (remifentanil) consumption, and postoperatively hemodynamics, pain scores (VAS), postoperative opioid [tramadol administered with a patient-controlled analgesia pump (PCA)] and, if necessary, rescue analgesic agent (non-steroidal antiinflammatory agent) consumption were monitored in the post anesthesia care unit (PACU), and at postoperative 6., 12. and 24.hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* ASA I and II
* Female
* Underwent mastectomy surgery
* Without local anesthetic allergy

Exclusion Criteria:

* Patients with ASA III and above
* Obesity (body mass index >30)
* Psychotropic drug use
* Bleeding diathesis
* Local anesthetic allergy
* Chest wall deformity
* Infection at the injection site
* Chronic analgesic usage

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Pain in the postoperative period was evaluated using the VAS score. | 24 hours
  The researchers investigate whether postoperative pain increases or decreases, using the VAS score at the postoperative anesthesia care unit, at postoperative 6 hours, 12 hours, and 24 hours.

SECONDARY OUTCOMES:
Incorporating the use of AI applications reduces the time required to block. | During the procedure.
  This software finds the image, implements the block quickly, and spends less time.

CONTACTS AND LOCATIONS:
Overall Officials: Elvin Kesimci, Study Director — Baskent University; Çağla Yazar, Principal Investigator — Baskent University
Locations (1):
- Çağla Yazar, MD, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Momenimovahed Z, Salehiniya H. Epidemiological characteristics of and risk factors for breast cancer in the world. Breast Cancer (Dove Med Press). 2019 Apr 10;11:151-164. doi: 10.2147/BCTT.S176070. eCollection 2019. PMID 31040712
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Bartakke DAA, Varma DMK. Analgesia for breast surgery - A Brief Overview. Medicine. 2019;7.
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Background] Bakeer AH, Kamel KM, Abdelgalil AS, Ghoneim AA, Abouel Soud AH, Hassan ME. Modified Pectoral Nerve Block versus Serratus Block for Analgesia Following Modified Radical Mastectomy: A Randomized Controlled Trial. J Pain Res. 2020 Jul 14;13:1769-1775. doi: 10.2147/JPR.S252539. eCollection 2020. PMID 32765052
- [Background] Karaca O, Pinar HU, Arpaci E, Dogan R, Cok OY, Ahiskalioglu A. The efficacy of ultrasound-guided type-I and type-II pectoral nerve blocks for postoperative analgesia after breast augmentation: A prospective, randomised study. Anaesth Crit Care Pain Med. 2019 Feb;38(1):47-52. doi: 10.1016/j.accpm.2018.03.009. Epub 2018 Apr 5. PMID 29627431
- [Background] la Grange P, Foster PA, Pretorius LK. Application of the Doppler ultrasound bloodflow detector in supraclavicular brachial plexus block. Br J Anaesth. 1978 Sep;50(9):965-7. doi: 10.1093/bja/50.9.965. PMID 708565
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Kuş A. Pektoral blok derleme. Türkiye Klinikleri Anesteziyoloji Reanimasyon - Özel Konular. 2015;8(3):74-7.
- [Background] Sites BD, Chan VW, Neal JM, Weller R, Grau T, Koscielniak-Nielsen ZJ, Ivani G; American Society of Regional Anesthesia and Pain Medicine; European Society Of Regional Anaesthesia and Pain Therapy Joint Committee. The American Society of Regional Anesthesia and Pain Medicine and the European Society Of Regional Anaesthesia and Pain Therapy Joint Committee recommendations for education and training in ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):40-6. doi: 10.1097/AAP.0b013e3181926779. PMID 19258987
- [Background] Akkus Z, Cai J, Boonrod A, Zeinoddini A, Weston AD, Philbrick KA, Erickson BJ. A Survey of Deep-Learning Applications in Ultrasound: Artificial Intelligence-Powered Ultrasound for Improving Clinical Workflow. J Am Coll Radiol. 2019 Sep;16(9 Pt B):1318-1328. doi: 10.1016/j.jacr.2019.06.004. PMID 31492410
- [Background] Bowness J, Varsou O, Turbitt L, Burkett-St Laurent D. Identifying anatomical structures on ultrasound: assistive artificial intelligence in ultrasound-guided regional anesthesia. Clin Anat. 2021 Jul;34(5):802-809. doi: 10.1002/ca.23742. Epub 2021 May 11. PMID 33904628
- [Background] Gungor I, Gunaydin B, Oktar SO, M Buyukgebiz B, Bagcaz S, Ozdemir MG, Inan G. A real-time anatomy identification via tool based on artificial intelligence for ultrasound-guided peripheral nerve block procedures: an accuracy study. J Anesth. 2021 Aug;35(4):591-594. doi: 10.1007/s00540-021-02947-3. Epub 2021 May 19. PMID 34008072
- [Background] Bowness J, El-Boghdadly K, Burckett-St Laurent D. Artificial intelligence for image interpretation in ultrasound-guided regional anaesthesia. Anaesthesia. 2021 May;76(5):602-607. doi: 10.1111/anae.15212. Epub 2020 Jul 29. No abstract available. PMID 32726498
- [Background] FitzGerald S, Odor PM, Barron A, Pawa A. Breast surgery and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2019 Mar;33(1):95-110. doi: 10.1016/j.bpa.2019.03.003. Epub 2019 Apr 6. PMID 31272657
- [Background] Hadzic A. Hadzic's Textbook of Regional Anesthesia and Acute Pain Management. 2nd edition. New York: McGraw Hill / Medical; 2017. 1536 p.
- [Background] Jacobs A, Lemoine A, Joshi GP, Van de Velde M, Bonnet F; PROSPECT Working Group collaborators#. PROSPECT guideline for oncological breast surgery: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2020 May;75(5):664-673. doi: 10.1111/anae.14964. Epub 2020 Jan 26. PMID 31984479
- [Background] Helander EM, Webb MP, Kendrick J, Montet T, Kaye AJ, Cornett EM, Kaye AD. PECS, serratus plane, erector spinae, and paravertebral blocks: A comprehensive review. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):573-581. doi: 10.1016/j.bpa.2019.07.003. Epub 2019 Jul 17. PMID 31791572
- [Background] Elsharkawy H, Pawa A, Mariano ER. Interfascial Plane Blocks: Back to Basics. Reg Anesth Pain Med. 2018 May;43(4):341-346. doi: 10.1097/AAP.0000000000000750. PMID 29561295
- [Background] Warfield DJ Jr, Barre S, Adhikary SD. Current understanding of the fascial plane blocks for analgesia of the chest wall: techniques and indications update for 2020. Curr Opin Anaesthesiol. 2020 Oct;33(5):692-697. doi: 10.1097/ACO.0000000000000909. PMID 32826623
- [Background] Lopez-Rincon RM, Hendrix JM, Kumar V. Ultrasound-Guided Intercostal Nerve Block. 2023 Jul 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK555900/ PMID 32310360
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Hinchcliff KM, Hylton JR, Orbay H, Wong MS. Intraoperative Placement of Pectoral Nerve Block Catheters: Description of a Novel Technique and Review of the Literature. Ann Plast Surg. 2017 May;78(5 Suppl 4):S189-S193. doi: 10.1097/SAP.0000000000000954. PMID 28118226
- [Background] Khemka R, Chakraborty A. Ultrasound-guided modified serratus anterior plane block for perioperative analgesia in breast oncoplastic surgery: A case series. Indian J Anaesth. 2019 Mar;63(3):231-234. doi: 10.4103/ija.IJA_752_18. PMID 30988539
- [Background] Afonso AM, Newman MI, Seeley N, Hutchins J, Smith KL, Mena G, Selber JC, Saint-Cyr MH, Gadsden JC. Multimodal Analgesia in Breast Surgical Procedures: Technical and Pharmacological Considerations for Liposomal Bupivacaine Use. Plast Reconstr Surg Glob Open. 2017 Sep 15;5(9):e1480. doi: 10.1097/GOX.0000000000001480. eCollection 2017 Sep. PMID 29062649
- [Background] Maheshwari K, Cywinski JB, Papay F, Khanna AK, Mathur P. Artificial Intelligence for Perioperative Medicine: Perioperative Intelligence. Anesth Analg. 2023 Apr 1;136(4):637-645. doi: 10.1213/ANE.0000000000005952. Epub 2023 Mar 16. PMID 35203086
- [Background] Hashimoto DA, Rosman G, Rus D, Meireles OR. Artificial Intelligence in Surgery: Promises and Perils. Ann Surg. 2018 Jul;268(1):70-76. doi: 10.1097/SLA.0000000000002693. PMID 29389679
- [Background] Nathan N. Perioperative Artificial Intelligence. Anesth Analg. 2023 Apr 1;136(4):636. doi: 10.1213/ANE.0000000000006427. Epub 2023 Mar 16. No abstract available. PMID 36928148
- [Background] Morse J, Terrasini N, Wehbe M, Philippona C, Zaouter C, Cyr S, Hemmerling TM. Comparison of success rates, learning curves, and inter-subject performance variability of robot-assisted and manual ultrasound-guided nerve block needle guidance in simulation. Br J Anaesth. 2014 Jun;112(6):1092-7. doi: 10.1093/bja/aet440. Epub 2014 Jan 23. PMID 24464610
- [Background] Bowness JS, El-Boghdadly K, Woodworth G, Noble JA, Higham H, Burckett-St Laurent D. Exploring the utility of assistive artificial intelligence for ultrasound scanning in regional anesthesia. Reg Anesth Pain Med. 2022 Jun;47(6):375-379. doi: 10.1136/rapm-2021-103368. Epub 2022 Jan 28. PMID 35091395
- [Background] Szamborski M, Janc J, Rosinczuk J, Janc JJ, Lesnik P, Lysenko L. Use of Ultrasound-Guided Interfascial Plane Blocks in Anterior and Lateral Thoracic Wall Region as Safe Method for Patient Anesthesia and Analgesia: Review of Techniques and Approaches during COVID-19 Pandemic. Int J Environ Res Public Health. 2022 Jul 17;19(14):8696. doi: 10.3390/ijerph19148696. PMID 35886547
- [Background] Kumar S, Goel D, Sharma SK, Ahmad S, Dwivedi P, Deo N, Rani R. A randomised controlled study of the post-operative analgesic efficacy of ultrasound-guided pectoral nerve block in the first 24 h after modified radical mastectomy. Indian J Anaesth. 2018 Jun;62(6):436-442. doi: 10.4103/ija.IJA_523_17. PMID 29962525
- [Background] Jindal R, Meena S, Bhati S, Patel P, Gulati C, Singh S. Postoperative Analgesic Efficacy of Intraoperative Pectoral Nerve Block for Modified Radical Mastectomy: a Double-Blind Prospective Randomised Interventional Study. Indian J Surg Oncol. 2023 Mar;14(1):215-221. doi: 10.1007/s13193-022-01680-x. Epub 2022 Nov 14. PMID 36891452
- [Background] Cesur S, Aksu C, Guler SA, Kus A. Modified pectoral nerve block versus bi-level erector spinae plane block for postoperative analgesia after radical mastectomy surgery: a prospective, randomized, controlled trial. Korean J Anesthesiol. 2023 Aug;76(4):317-325. doi: 10.4097/kja.22188. Epub 2023 Mar 14. PMID 36916186
- [Background] Kocer Tulgar Y, Tulgar S, Guven Kose S, Kose HC, Cevik Nasirlier G, Dogan M, Thomas DT. Anesthesiologists' Perspective on the Use of Artificial Intelligence in Ultrasound-Guided Regional Anaesthesia in Terms of Medical Ethics and Medical Education: A Survey Study. Eurasian J Med. 2023 Jun;55(2):146-151. doi: 10.5152/eurasianjmed.2023.22254. PMID 37161553